CLINICAL TRIAL: NCT02851433
Title: Evaluate the Protective Effect of Conditioning With Sevoflurane Versus Propofol on the Myocardium in Scheduled Aortic Valve Replacement Surgery
Brief Title: Evaluate the Protective Effect of Conditioning With Sevoflurane on the Myocardium
Acronym: SUPRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JAUDON-FAIVRE 2014
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Cardiac Surgery
MeSH Terms: interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Sevoflurane Group (Experimental)
  Interventions: Drug: total anaesthesia and postoperative inhaled sedation with Sevoflurane
- Propofol Group (Active Comparator)
  Interventions: Drug: total intravenous anaesthesia with Propofol.

INTERVENTIONS:
Drug: total anaesthesia and postoperative inhaled sedation with Sevoflurane
  Arms: Sevoflurane Group
Drug: total intravenous anaesthesia with Propofol.
  Arms: Propofol Group

SUMMARY:
Heart surgery is a considerable source of stress for the myocardium that must be minimized.

Troponin Ic is a reliable marker to determine the level of this myocardial stress.

Studies have shown that post-conditioning with AVH has a protective effect on the myocardium, if the treatment is initiated at the start of the ischemia.

The aim of this study is to evaluate the protective effect on the myocardium (by measuring troponin levels) of the association of pre-conditioning and post-conditioning with Sevoflurane (AVH) sedation administered during and after scheduled surgery for valve replacement, via sternotomy or thoracotomy compared with total intravenous anaesthesia with Propofol.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided informed written consent.
* Aortic valve replacement via sternotomy or thoracotomy, under Cardiopulmonary bypass (CPB).
* Anterograde cardioplegia with cold blood

Exclusion Criteria:

* Adults under guardianship.
* Patients without national health insurance cover.
* Epileptics.
* Heart grafted patients.
* Patients under 18 years and pregnant or beast-feeding women.
* Aortic dissections and vascular surgery.
* Contra-indications to treatment with Sevoflurane: hypersensitivity to halogen-based anaesthetic agents, myopathy, personal or family history of malignant hyperthermia, hyper-eosinophilia, liver disease, icterus or unexplained fever after anaesthesia with a halogen-based anaesthetic agent
* Contra-indications to treatment with Propofol: known hypersensitivity to propofol or one of the constituents of the specific form used, hypersensitivity to peanuts or soja.
* pre-operative LVEF<35%.
* Coronary artery bypass graft alone or associated.
* Mitral valve replacements.
* Warm cardioplegia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-10-14 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2017-09-04 (Actual)

PRIMARY OUTCOMES:
Levels of troponin | Change at Hour 6, Hour 12, Hour 24, Hour 48 compared with baseline level

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Guinot PG, Ellouze O, Grosjean S, Berthoud V, Constandache T, Radhouani M, Anciaux JB, Aho-Glele S, Morgant MC, Girard C, Nguyen M, Bouhemad B. Anaesthesia and ICU sedation with sevoflurane do not reduce myocardial injury in patients undergoing cardiac surgery: A randomized prospective study. Medicine (Baltimore). 2020 Dec 11;99(50):e23253. doi: 10.1097/MD.0000000000023253. PMID 33327246